CLINICAL TRIAL: NCT01566955
Title: Feasability of Transgastric Adnexectomy
Brief Title: Feasability Study of Removing the Ovaries and Fallopian Tubes
Acronym: TG-Adnex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dr. med. Amadeus Hornemann, MPH, Dr. Amadeus Hornemann, MPH, PhD, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMM-Mannheim
Record Dates: First submitted 2012-03-22; First posted 2012-03-30 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Ovarian Diseases
Keywords: transgastric; NOTES; Gastrotomy; BRCA 1/2
MeSH Terms: conditions — Ovarian Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- transgastric adnexectomy (Experimental): patients are operated transgastric
  Interventions: Procedure: transgastric adnexectomy

INTERVENTIONS:
Procedure: transgastric adnexectomy — adnexectomy transgastrically with transvaginal support
  Other Names: NOTES; Pure NOTES

SUMMARY:
The main reason for this trial is to show the feasibility of removing the ovarien and fallopian tubes through the gaster (transgastric adnexectomy). The background for it is to look for more indications of scarless surgery and we will show that the transgastric adnexectomy can be performed in an easy way. It is necessary that there is an indication for removing the ovaries and fallopian tubes and if the patient agree we will do it instead of through the belly through the gaster and maybe with an additional inzision in the vagina. All patients with indication for adnexectomy are potential candidates.

DETAILED DESCRIPTION:
We will show the feasibility for transgastric adnexectomy in 10 patients. Patients for participating in the study suffer of benign adnexal deseases and there is an indication for removing them for diagnostic, prophylactic or therapeutic reasons. A flexible gastric scope is put transgastric into the abdomen, developing an pneumoperitoneum and removing the adnexes with a monopolar knife. The adnexes then are put out of the abdomen either transvaginally after colpotomy or even transgastric. We already performed an appendectomy in 24 patients and were able to show the feasibility in acute infectios situations.

ELIGIBILITY:
Inclusion Criteria:

* Indication for adnexectomy, agreement to take part in the study

Exclusion Criteria:

* No agreement in the trial; patients younger than 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with conversion to laparoscopy or laparotomy | 12 months
  With the trial we want to demonstrate that the transgastric adnexectomy is possible. We will document the number of patients in which we have to change the transgastric to a laparoscopic or laparotomic operation.

SECONDARY OUTCOMES:
postoperative well being | 6 weeks and 6 months
  Postoperative well being after 6 weeks and after 6 months (standardized questionaire of our hospital)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Suetterlin, MD; PhD, Study Chair — University of Heidelberg, University Medical Center Mannheim Department of Obstetric and Gynaecology
Locations (1):
- University Medical Center Mannheim, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Hornemann A, Suetterlin M, Trunk MJ, Gerhardt A, Kaehler G. Pure natural orifice transluminal endoscopic surgery (NOTES) involving peroral endoscopic salpingo-oophorectomy (POESY). Int J Gynaecol Obstet. 2014 Apr;125(1):86-8. doi: 10.1016/j.ijgo.2013.08.024. Epub 2014 Jan 2. PMID 24434232